CLINICAL TRIAL: NCT00372957
Title: PK/PD Study of GW823093 in Japanese Subjects With T2DM: A Single-blind, Placebo Controlled, Randomized, Multi-dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GW823093C Administered Orally for 7 Days in Japanese Subjects With Type 2 Diabetes
Brief Title: Study Of GW823093 In Japanese Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: DPB106653
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacodynamics; Diabetes; pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

ARMS (3):
- Placebo (Placebo Comparator): Participants received two capsules of matching placebo orally once daily in the morning with 150 milliliter (mL) of water at least 15 minutes prior to breakfast for 7 Days.
  Interventions: Drug: GW823093 placebo capsule
- GW823093C 15 mg (Experimental): Participants received one 15 milligrams (mg) of GW823093C capsule and one placebo capsule orally once daily in the morning with 150 mL of water at least 15 minutes prior to breakfast for 7 Days.
  Interventions: Drug: GW823093 15mg; Drug: GW823093 placebo capsule
- GW823093C 30 mg (Experimental): Participants received 30 mg (2x15 mg) of GW823093C capsules orally once daily in the morning with 150 mL of water at least 15 minutes prior to breakfast for 7 Days.
  Interventions: Drug: GW823093 30mg

INTERVENTIONS:
Drug: GW823093 15mg — White opaque capsule containing 15mg of GW823093 as free base
  Other Names: GW823093
  Arms: GW823093C 15 mg
Drug: GW823093 placebo capsule — Matching placebo of GW823093 capsule or 15mg capsule
  Arms: GW823093C 15 mg; Placebo
Drug: GW823093 30mg — White opaque capsule containing 15mg of GW823093 as free base
  Arms: GW823093C 30 mg

SUMMARY:
To investigate the preliminary pharmacokinetics, pharmacodynamics, safety and tolerability of GW823093 at doses of 15mg and 30mg given once daily for 7 days in Japanese Type 2 diabetes mellitus (T2DM) patients.

ELIGIBILITY:
Inclusion criteria:

* T2DM diagnosed at least 3 months prior to Screening and fasting plasma glucose (FPG) level <280mg/dL at the Screening visit.
* Concurrent T2DM therapy: Must be diet controlled - OR - not taking more than 2 oral anti-diabetic agents, and willing to withdraw from these treatments 2 weeks prior to the first dosing.

Exclusion criteria:

* Must not have any other major illness other than diabetes

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03-22 (Actual); Primary Completion 2006-06-28 (Actual); Study Completion 2006-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across two centers in Japan from 22 March 2006 to 28 June 2006.
Pre-assignment Details: A total of 30 participants were randomized in the study. After screening, participants were washed off of diabetes medications for two weeks prior to the first dose of study medication.
Period: Overall Study
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received two capsules of matching placebo orally once daily in the morning with 150 mL of water at least 15 minutes prior to breakfast for 7 Days.
- GW823093C 15 mg: Participants received one 15 mg of GW823093C capsule and one placebo capsule orally once daily in the morning with 150 mL of water at least 15 minutes prior to breakfast for 7 Days.
- Total: Total of all reporting groups
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Customized [Count of Participants; unit: Participants]
  20 to 64 Years | 10 | 10 | 10 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 8 | 9 | 8 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 10 | 10 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Standard Pharmacokinetic (PK) Parameter: Maximum Observed Plasma Drug Concentration (Cmax)
Description: PK parameters were calculated using data at the actual time of blood collection. Cmax was determined from plasma concentration-time data, using standard model independent methods.
Time Frame: Day 1 (at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 hours [hr]), Day 2 (0 hr) and Day 7 (0, 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hr)
Population: PK Parameter Population comprised of all participants who received an active dose of GW823093C and for whom PK data was collected.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter (ng/mL)
Arm/Group | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10
Nanograms per milliliter (ng/mL)
  Day 1 | 238.166 [183.730 to 308.731] | 419.937 [358.461 to 491.957]
  Day 7 | 262.523 [209.416 to 329.097] | 534.888 [486.074 to 588.604]

2. Primary Outcome: Standard PK Parameter: Time at Which Cmax Was Observed (Tmax)
Description: PK parameters were calculated using data at the actual time of blood collection. Tmax was determined from plasma concentration-time data, using standard model independent methods.
Time Frame: Day 1 (at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 hr), Day 2 (0 hr) and Day 7 (0, 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hr)
Population: PK Parameter Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10
Hour
  Tmax, Day 1 | 2.50 [0.5 to 4.0] | 3.50 [0.5 to 6.0]
  Tmax, Day 7 | 3.00 [0.5 to 4.0] | 2.00 [0.5 to 4.0]

3. Primary Outcome: Standard PK Parameter: Half Life of Terminal Elimination Phase (t1/2)
Description: PK parameters were calculated using data at the actual time of blood collection. T1/2 was determined from plasma concentration-time data, using standard model independent methods.
Time Frame: Day 1 (at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 hr), Day 2 (0 hr) and Day 7 (0, 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hr)
Population: PK Parameter Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Hour
Arm/Group | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10
Hour
  Day 1 | 6.662 [5.884 to 7.543] | 8.788 [8.094 to 9.541]
  Day 7 | 7.127 [6.372 to 7.971] | 9.648 [8.674 to 10.731]

4. Primary Outcome: Standard PK Parameter: Area Under the Plasma Drug Concentration Versus Time Curve Extrapolated to Infinity (AUC[0-inf]), AUC From 0 to the Last Measurable Concentration (AUC[0-t])
Description: PK parameters were calculated using data at the actual time of blood collection. AUC[0-inf] and AUC[0-t] was determined from plasma concentration-time data, using standard model independent methods.
Time Frame: Day 1 (at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 hr), Day 2 (0 hr) and Day 7 (0, 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hr)
Population: PK Parameter Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Hr.ng/mL
Arm/Group | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10
Hr.ng/mL
  AUC(0-t), Day 1 | 2261.076 [1944.959 to 2628.572] | 4800.677 [4451.224 to 5177.565]
  AUC(0-t), Day 7 | 2545.651 [2155.396 to 3006.567] | 6129.987 [5801.218 to 6477.387]
  AUC(0-inf), Day 1 | 2508.608 [2114.506 to 2976.163] | 5786.001 [5449.326 to 6143.477]
  AUC(0-inf), Day 7 | 2870.716 [2374.654 to 3470.405] | 7562.008 [7132.565 to 8017.307]

5. Primary Outcome: Standard PK Parameter: Percentage of AUC(0-inf) Obtained by Extrapolation (%AUCex)
Description: PK parameters were calculated using data at the actual time of blood collection. %AUCex was determined from plasma concentration-time data, using standard model independent methods.
Time Frame: Day 1 (at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 hr), Day 2 (0 hr) and Day 7 (0, 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hr)
Population: PK Parameter Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of AUCex
Arm/Group | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10
Percentage of AUCex
  Day 1 | 9.029 [6.625 to 12.305] | 16.645 [14.331 to 19.333]
  Day 7 | 10.704 [8.425 to 13.601] | 18.442 [15.817 to 21.503]

6. Primary Outcome: Standard PK Parameter: Constant Rate of Elimination (lambda_z)
Description: PK parameters were calculated using data at the actual time of blood collection. Lambda_z was determined from plasma concentration-time data, using standard model independent methods.
Time Frame: Day 1 (at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 hr), Day 2 (0 hr) and Day 7 (0, 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hr)
Population: PK Parameter Population.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/hr
Arm/Group | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10
1/hr
  Day 1 | 0.10403 [0.09188 to 0.11779] | 0.07887 [0.07266 to 0.08562]
  Day 7 | 0.09727 [0.08697 to 0.10879] | 0.07184 [0.06458 to 0.07992]

7. Primary Outcome: Standard PK Parameter: Total Clearance (CL/F)
Description: PK parameters were calculated using data at the actual time of blood collection. CL/F was determined from plasma concentration-time data, using standard model independent methods.
Time Frame: Day 1 (at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 hr), Day 2 (0 hr) and Day 7 (0, 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hr)
Population: PK Parameter Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter per hour (L/hr)
Arm/Group | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10
Liter per hour (L/hr)
  Day 1 | 5.979 [5.040 to 7.094] | 5.185 [4.883 to 5.505]
  Day 7 | 5.225 [4.322 to 6.317] | 3.967 [3.742 to 4.206]

8. Primary Outcome: Standard PK Parameter: Apparent Volume of Distribution (Vz/F)
Description: PK parameters were calculated using data at the actual time of blood collection. Vz/F was determined from plasma concentration-time data, using standard model independent methods.
Time Frame: Day 1 (at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 hr), Day 2 (0 hr) and Day 7 (0, 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hr)
Population: PK Parameter Population.
Measure: Geometric Mean (95% Confidence Interval); unit: L
Arm/Group | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10
L
  Day 1 | 57.470 [51.466 to 64.175] | 65.735 [58.465 to 73.910]
  Day 7 | 53.724 [48.155 to 59.938] | 55.221 [50.088 to 60.881]

9. Primary Outcome: Standard PK Parameter: R[Cmax], Extent of Accumulation (Ro), Steady State Accumulation Ratio (Rs)
Description: PK parameters were calculated using data at the actual time of blood collection. R[Cmax], Ro and Rs were determined from plasma concentration-time data, using standard model independent methods. R[Cmax] = Cmax (Day 7)/Cmax (Day 1), Ro = AUC(0-tau) (Day 7)/ AUC(0-tau) (Day 1) and Rs = AUC(0-tau) (Day 7)/ AUC(0-inf) (Day 1).
Time Frame: Day 1 (at 0, 1, 1.5, 2, 3, 4, 6, 8, 12 hr), Day 2 (0 hr) and Day 7 (0, 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 hr)
Population: PK Parameter Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10
Ratio
  R[Cmax] | 1.102 [0.946 to 1.284] | 1.274 [1.110 to 1.461]
  Ro | 1.126 [1.082 to 1.171] | 1.277 [1.183 to 1.379]
  Rs | 1.015 [0.987 to 1.044] | 1.059 [0.988 to 1.136]

10. Primary Outcome: Percent Dipeptidyl-peptidase IV (DPP-IV) Inhibition by Dose (Day 7)
Description: For analysis of DPP-IV activity, approximately 2 mL of whole blood was collected into a vacuum tube containing ethylenediamine tetraacetic acid (EDTA2K) and centrifuged at approximately 4 degree Celsius, at approximately 2500 revolution per minute (rpm) for 15 minutes. Samples were stored in a freezer at -70 degree Celsius or lower. DPP-IV inhibition was estimated by using the percent change from pre-dose of DPP-IV activity. DPP-IV inhibition was done at pre-dose, 0.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr and 24 hr.
Time Frame: Day 7
Population: Pharmacodynamic (PD) Parameter Population comprised of all participants who received study medication (active or placebo) and for whom PD data was available.
Measure: Number; unit: Percent inhibition
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10 | 10
Percent inhibition
  Pre-dose | 0.000 | 69.565 | 88.854
  0.5hr | 2.273 | 83.612 | 88.854
  1hr | -1.724 | 91.107 | 91.033
  1.5hr | 0.000 | 91.304 | 91.033
  2hr | -1.724 | 91.304 | 92.593
  3hr | -2.273 | 91.304 | 92.593
  4hr | -3.448 | 91.304 | 92.593
  6 hr | -5.721 | 91.107 | 91.609
  8 hr | -9.091 | 91.107 | 92.593
  12 hr | -9.091 | 91.107 | 91.033
  24 hr | -4.105 | 68.783 | 88.562

11. Primary Outcome: DPP-IV Activity Weighted Mean AUCs at Baseline (Day -1) and Day 7
Description: For analysis of DPP-IV activity, approximately 2 mL of whole blood was collected into a vacuum tube containing EDTA2K and centrifuged at approximately 4 degree Celsius, at approximately 2500 rpm for 15 minutes. Samples were stored in a freezer at -70 degree Celsius or lower. Double-delta represented active treatment within participant change from Baseline summarized across participants, subtracted from placebo within participant change from Baseline summarized across participants. AUC with respect to these time interval was calculated using linear trapezoidal rule by sum of the areas between each chronological pair of assessments (using observed times). Weighted mean was then determined by dividing AUC by observed length of collection interval (time of last assessment - time of first assessment in hr). Double-delta analysis has been presented in analysis. Unit of measure: Nano mole per minute per milliliter (nmol/min/mL).
Time Frame: Baseline (Day -1) and Day 7
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: nmol/min/mL
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10 | 10
nmol/min/mL
  AUC(0-12 hr), Day -1 | 2.34 (0.38) | 2.43 (0.25) | 2.41 (0.70)
  AUC(0-12 hr), Day 7 | 2.35 (0.35) | 0.27 (0.08) | 0.21 (0.02)
  AUC(0-24 hr), Day -1 | 2.35 (0.38) | 2.44 (0.28) | 2.42 (0.71)
  AUC(0-24 hr), Day 7 | 2.34 (0.32) | 0.37 (0.12) | 0.23 (0.06)
Statistical Analysis 1: Comparison: Placebo vs GW823093C 15 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -2.10, 95% CI 2-sided [-2.28 to -1.93] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 2: Comparison: Placebo vs GW823093C 30 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-2.33 to -1.98] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg
Statistical Analysis 3: Comparison: Placebo vs GW823093C 15 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.15 to -1.82] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 4: Comparison: Placebo vs GW823093C 30 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -2.12, 95% CI 2-sided [-2.28 to -1.95] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg

12. Primary Outcome: Active Glucagon-like Peptide-1 (GLP-1) Weighted Mean AUCs at Baseline (Day -1) and Day 7
Description: For the analysis of active GLP-1 concentrations, approximately 3 mL of whole blood was collected into a vacuum tube containing DPP-IV inhibitor, and then centrifuged in a refrigerated centrifuge at approximately 4 degree Celsius, at approximately 2500 rpm for 15 minutes. Samples were stored in a freezer at -70 degree Celsius or lower. Double-delta represented the active treatment within participant change from Baseline summarized across participants, subtracted from placebo within participant change from Baseline summarized across participants. AUC with respect to these time interval was calculated using linear trapezoidal rule by sum of the areas between each chronological pair of assessments (using observed times). Weighted mean was then determined by dividing AUC by observed length of collection interval (time of last assessment - time of first assessment in hr). Double-delta analysis for weighted mean AUCs has been presented in the statistical analysis section.
Time Frame: Baseline (Day -1) and Day 7
Population: PD Parameter Population.
Measure: Mean (Standard Deviation); unit: Picomole (pM)
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10 | 10
Picomole (pM)
  AUC(0-12 hr), Day -1 | 4.64 (3.68) | 3.21 (1.06) | 5.48 (3.04)
  AUC(0-12 hr), Day 7 | 4.74 (3.80) | 7.19 (2.46) | 10.79 (3.32)
  AUC(0-24 hr), Day -1 | 4.25 (3.34) | 2.77 (0.80) | 4.99 (2.64)
  AUC(0-24 hr), Day 7 | 4.65 (3.54) | 6.37 (2.22) | 9.81 (2.77)
Statistical Analysis 1: Comparison: Placebo vs GW823093C 15 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 3.87, 95% CI 2-sided [2.33 to 5.41] — he point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 2: Comparison: Placebo vs GW823093C 30 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 5.21, 95% CI 2-sided [3.70 to 6.73] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg
Statistical Analysis 3: Comparison: Placebo vs GW823093C 15 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 3.22, 95% CI 2-sided [1.90 to 4.54] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 4: Comparison: Placebo vs GW823093C 30 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 4.39, 95% CI 2-sided [3.10 to 5.68] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg

13. Primary Outcome: Insulin Weighted Mean AUCs at Baseline (Day -1) and Day 7
Description: For the analysis of plasma insulin, approximately 2 mL of whole blood was collected into a vacuum tube containing EDTA2Na, and then centrifuged in a refrigerated centrifuge at approximately 4 degree Celsius, at approximately 2500 rpm for 15 minutes. Samples were stored in a freezer at -70 degree Celsius or lower. Double-delta represented the active treatment within participant change from Baseline summarized across participants, subtracted from placebo within participant change from Baseline summarized across participants. AUC with respect to these time interval was calculated using linear trapezoidal rule by sum of the areas between each chronological pair of assessments (using observed times). Weighted mean was then determined by dividing AUC by observed length of collection interval (time of last assessment - time of first assessment in hr). Double-delta analysis for weighted mean AUCs has been presented in the statistical analysis section.
Time Frame: Baseline (Day -1) and Day 7
Population: PD Parameter Population.
Measure: Mean (Standard Deviation); unit: Micro units per milliliter (µU/mL)
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10 | 10
Micro units per milliliter (µU/mL)
  AUC(0-12 hr), Day -1 | 17.35 (7.37) | 17.55 (7.72) | 21.28 (12.06)
  AUC(0-12 hr), Day 7 | 18.07 (9.28) | 16.70 (6.75) | 22.79 (11.95)
  AUC(0-24 hr), Day -1 | 16.60 (6.75) | 17.87 (7.68) | 21.72 (12.66)
  AUC(0-24 hr), Day 7 | 16.89 (7.73) | 16.64 (6.91) | 22.81 (11.90)
Statistical Analysis 1: Comparison: Placebo vs GW823093C 15 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -1.56, 95% CI 2-sided [-6.00 to 2.89] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 2: Comparison: Placebo vs GW823093C 30 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [-3.30 to 5.72] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg
Statistical Analysis 3: Comparison: Placebo vs GW823093C 15 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-5.20 to 2.50] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 4: Comparison: Placebo vs GW823093C 30 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [-2.47 to 5.43] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg

14. Primary Outcome: Glucagon Weighted Mean AUCs at Baseline (Day -1) and Day 7
Description: For the analysis of plasma glucagons concentrations, approximately 2 mL of whole blood was collected into a vacuum tube containing aprotinin, and then centrifuged in a refrigerated centrifuge at approximately 4 degree Celsius, at approximately 2500 rpm for 15 minutes. Samples were stored in a freezer at -70 degree Celsius or lower. Double-delta represented the active treatment within participant change from Baseline summarized across participants, subtracted from placebo within participant change from Baseline summarized across participants. AUC with respect to these time interval was calculated using linear trapezoidal rule by sum of the areas between each chronological pair of assessments (using observed times). Weighted mean was then determined by dividing AUC by observed length of collection interval (time of last assessment - time of first assessment in hr). Double-delta analysis for weighted mean AUCs has been presented in the statistical analysis section.
Time Frame: Baseline (Day -1) and Day 7
Population: PD Parameter Population.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter (pg/mL)
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10 | 10
Picogram per milliliter (pg/mL)
  AUC(0-12 hr), Day -1 | 113.1 (49.2) | 100.1 (14.9) | 125.1 (37.0)
  AUC(0-12 hr), Day 7 | 113.9 (34.4) | 97.3 (17.3) | 105.6 (27.2)
  AUC(0-24 hr), Day -1 | 114.7 (53.2) | 104.4 (16.9) | 129.0 (41.0)
  AUC(0-24 hr), Day 7 | 113.4 (32.5) | 97.0 (16.3) | 105.6 (24.3)
Statistical Analysis 1: Comparison: Placebo vs GW823093C 15 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -8.1, 95% CI 2-sided [-20.4 to 4.2] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 2: Comparison: Placebo vs GW823093C 30 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -16.2, 95% CI 2-sided [-28.4 to -3.9] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg
Statistical Analysis 3: Comparison: Placebo vs GW823093C 15 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -10.9, 95% CI 2-sided [-23.1 to 1.4] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 4: Comparison: Placebo vs GW823093C 30 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -15.6, 95% CI 2-sided [-27.9 to -3.3] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg

15. Primary Outcome: C-peptide Weighted Mean AUCs at Baseline (Day -1) and Day 7
Description: For the analysis of plasma C-peptide concentrations, approximately 2 mL of whole blood was collected into a vacuum tube containing EDTA2Na, and then centrifuged in a refrigerated centrifuge at approximately 4 degree Celsius, at approximately 2500 rpm for 15 minutes. Samples were stored in a freezer at -70 degree Celsius or lower. Double-delta represented the active treatment within participant change from Baseline summarized across participants, subtracted from placebo within participant change from Baseline summarized across participants. AUC with respect to these time interval was calculated using linear trapezoidal rule by sum of the areas between each chronological pair of assessments (using observed times). Weighted mean was then determined by dividing AUC by observed length of collection interval (time of last assessment - time of first assessment in hr). Double-delta analysis for weighted mean AUCs has been presented in the statistical analysis section.
Time Frame: Baseline (Day -1) and Day 7
Population: PD Parameter Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10 | 10
ng/mL
  AUC(0-12 hr), Day -1 | 4.29 (1.25) | 3.78 (1.54) | 4.73 (1.29)
  AUC(0-12 hr), Day 7 | 4.46 (1.20) | 4.31 (1.27) | 5.25 (1.83)
  AUC(0-24 hr), Day -1 | 3.88 (1.02) | 3.54 (1.41) | 4.40 (1.30)
  AUC(0-24 hr), Day 7 | 4.01 (0.90) | 4.07 (1.18) | 4.94 (1.72)
Statistical Analysis 1: Comparison: Placebo vs GW823093C 15 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.64 to 1.16] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 2: Comparison: Placebo vs GW823093C 30 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-0.47 to 1.32] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg
Statistical Analysis 3: Comparison: Placebo vs GW823093C 15 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.37 to 1.07] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 4: Comparison: Placebo vs GW823093C 30 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-0.24 to 1.21] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg

16. Primary Outcome: Glucose Weighted Mean AUCs at Baseline (Day -1) and Day 7
Description: For the analysis of plasma glucose concentrations, approximately 2 mL of whole blood was collected into a vacuum tube containing sodium fluoride, and then centrifuged in a refrigerated centrifuge at approximately 4 degree Celsius, at approximately 2500 rpm for 15 minutes. Samples were stored in a freezer at -70 degree Celsius or lower. Double-delta represented the active treatment within participant change from Baseline summarized across participants, subtracted from placebo within participant change from Baseline summarized across participants. AUC with respect to these time interval was calculated using linear trapezoidal rule by sum of the areas between each chronological pair of assessments (using observed times). Weighted mean was then determined by dividing AUC by observed length of collection interval (time of last assessment - time of first assessment in hr). Double-delta analysis for weighted mean AUCs has been presented in the statistical analysis section.
Time Frame: Baseline (Day -1) and Day 7
Population: PD Parameter Population.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10 | 10
Milligrams per deciliter (mg/dL)
  AUC(0-12 hr), Day -1 | 218.9 (69.5) | 233.8 (68.7) | 227.5 (64.1)
  AUC(0-12 hr), Day 7 | 210.0 (73.5) | 203.2 (52.5) | 208.6 (62.1)
  AUC(0-24 hr), Day -1 | 211.4 (66.0) | 221.6 (58.2) | 219.1 (51.6)
  AUC(0-24 hr), Day 7 | 201.1 (67.2) | 194.6 (45.5) | 202.0 (55.5)
Statistical Analysis 1: Comparison: Placebo vs GW823093C 15 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -19.9, 95% CI 2-sided [-40.7 to 0.9] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 2: Comparison: Placebo vs GW823093C 30 mg; AUC(0-12 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -9.0, 95% CI 2-sided [-29.8 to 11.7] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg
Statistical Analysis 3: Comparison: Placebo vs GW823093C 15 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -15.9, 95% CI 2-sided [-33.2 to 1.4] — The point estimate is the least square mean difference between placebo and GW 823093C 15 mg
Statistical Analysis 4: Comparison: Placebo vs GW823093C 30 mg; AUC(0-24 hr), Day 7; Test type: Superiority or Other; Double-delta analysis; Mean Difference (Final Values) = -6.2, 95% CI 2-sided [-23.4 to 11.1] — The point estimate is the least square mean difference between placebo and GW 823093C 30 mg

17. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is serious corresponding to those listed in above definition.
Time Frame: Up to post-study screen (Follow-up [7 days after the last dose of study medication])
Population: Safety Population comprised of all participants who received study medication (active or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Any AEs | 1 | 0 | 0
  Any SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected up to post-study screen (Follow-up [7 days after the last dose of study medication]).
Description: Safety Population was used for the analysis.
Arm/Group | Placebo | GW823093C 15 mg | GW823093C 30 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | GW823093C 15 mg (N=10) | GW823093C 30 mg (N=10)
Herpes zoster (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.